CLINICAL TRIAL: NCT02000921
Title: Models for Tobacco Productive Evaluation: Reduced Nicotine Content Cigarettes and Tobacco Switching Behaviors
Brief Title: Reduced Nicotine Content Cigarettes and Tobacco Switching Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2013NTLS012; U19CA157345 (NIH)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Tobacco Addiction; Dual Tobacco Use
Keywords: Cigarette Smoking; Very Low Nicotine Content cigarettes (VLNC); Dual Tobacco Use
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CN + combusted & non-combusted products (Experimental): Subjects will be asked to smoke the assigned conventional nicotine content (CN) cigarettes, instead of their normal brand, for 8 weeks and will also be given access to use other combusted and non-combusted tobacco and medicinal nicotine products during that time.
  Interventions: Other: Combusted Products; Other: Non-combusted products; Other: CN cigarettes
- VLNC + combusted & non-combusted products (Experimental): Subjects will be asked to smoke the assigned very low nicotine content (VLNC) cigarettes, instead of their normal brand, for 8 weeks and will also be given access to use other combusted and non-combusted tobacco and medicinal nicotine products during that time.
  Interventions: Other: VLNC cigarettes; Other: Combusted Products; Other: Non-combusted products
- VLNC with non-combusted products (Experimental): Subjects will be asked to smoke very low nicotine content (VLNC) cigarettes instead of their usual cigarettes for an 8 week period and will be given the opportunity to use non-combusted types of tobacco and medicinal tobacco products.
  Interventions: Other: VLNC cigarettes; Other: Non-combusted products

INTERVENTIONS:
Other: VLNC cigarettes — Modified risk tobacco product
  Other Names: Very Low Nicotine Content Cigarettes
  Arms: VLNC + combusted & non-combusted products; VLNC with non-combusted products
Other: Combusted Products — Options for combusted tobacco products include cigars, cigarillos, and little cigars, .
  Arms: CN + combusted & non-combusted products; VLNC + combusted & non-combusted products
Other: Non-combusted products — Options for non-combusted tobacco products include smokeless tobacco, novel snus products, e-cigarettes and medicinal nicotine.
Other: CN cigarettes — Experimental cigarettes with conventional nicotine content.
  Arms: CN + combusted & non-combusted products

SUMMARY:
The main focus of this study is to determine the use of nicotine-containing products across the three experimental conditions. Subjects will be monitored to determine their continued use of assigned cigarettes, switching to other combusted and/or non-combusted tobacco, or cessation of all tobacco containing products.

DETAILED DESCRIPTION:
This is a single site, single-blind, randomized trial with three experimental conditions tested for a period of 8 weeks: 1) Very low nicotine content (VLNC) cigarettes (0.07 nicotine yield) with access to combusted (except cigarettes) and non-combusted tobacco and medicinal nicotine products; 2) VLNC cigarettes with access to only non-combusted tobacco and medicinal nicotine products; and 3) conventional nicotine (CN) content experimental cigarettes (0.8 mg nicotine) with access to combusted and non-combusted products. This study will examine the use of nicotine-containing products across the three experimental conditions. Subjects will be monitored to determine their continued use of assigned cigarettes, switching to other combusted (e.g., little cigars, large cigars, pipes) and/or non-combusted tobacco products (e.g., conventional smokeless tobacco, snus for smokers, dissolvables, e-cigarettes, medicinal nicotine), or cessation of all tobacco containing products. Toxicant exposure across the three conditions will also be examined.

Eligible subjects will be provided very low nicotine content cigarettes and are told to use the product ad lib for 8 weeks. Subjects will complete questionnaires on demographics, smoking and health history, drug and alcohol use history, mood and perceptions of the study tobacco product. Biomarker samples will be analyzed for exposure levels of nicotine and tobacco-related toxicants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are at least 18 years of age with a history of regular smoking for at least 1 year and no serious quit attempts in the last 3 months
* No unstable and significant medical or psychiatric conditions, including lack of stabilization of medications.
* Subject has provided written informed consent to participate in the study

Exclusion Criteria:

* Regular use of tobacco products (including e-cigarettes) other than cigarettes
* Regular use of nicotine replacement or other tobacco cessation products for purpose of quitting.
* Pregnant or breastfeeding (due to toxic effects from tobacco products).
* Planned quit date within the next two months.
* Does not have a way that the research team can communicate with them by phone or e-mail.
* Not able to read and write English well enough to complete study activities without translation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Tobacco Research Program, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hatsukami DK, Luo X, Dick L, Kangkum M, Allen SS, Murphy SE, Hecht SS, Shields PG, al'Absi M. Reduced nicotine content cigarettes and use of alternative nicotine products: exploratory trial. Addiction. 2017 Jan;112(1):156-167. doi: 10.1111/add.13603. Epub 2016 Nov 2. PMID 27614097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CN + Combusted & Non-combusted Products | VLNC + Combusted & Non-combusted Products | VLNC With Non-combusted Products
Started | 27 | 53 | 56
Completed | 22 | 37 | 46
Not Completed | 5 | 16 | 10
Not completed — Withdrawal by Subject | 3 | 10 | 5
Not completed — Lost to Follow-up | 2 | 4 | 5
Not completed — Physician Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CN + Combusted & Non-combusted Products | VLNC + Combusted & Non-combusted Products | VLNC With Non-combusted Products | Total
Number analyzed (Participants) | 27 | 53 | 56 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 3 | 3
  Between 18 and 65 years | 26 | 48 | 49 | 123
  >=65 years | 1 | 5 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (14) | 44 (15) | 45 (15) | 44 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 29 | 29 | 69
  Male | 16 | 24 | 27 | 67
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 53 | 56 | 136

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Using Alternative Products
Description: The primary aim of the study is to determine the rate of use of alternative nicotine-containing products across the three experimental conditions.
Time Frame: 8 week intervetnion period
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | CN + Combusted & Non-combusted Products | VLNC + Combusted & Non-combusted Products | VLNC With Non-combusted Products
Number analyzed (Participants) | 27 | 53 | 56
Number of days | 14 (17) | 26 (19) | 20 (19)

2. Primary Outcome: Number of Combusted Products Smoked
Description: Number of combusted products smoked per day during the last two weeks of the intervention period.
Time Frame: At weeks 6-8 (last two weeks of intervention period)
Measure: Mean (Standard Deviation); unit: combuster products per day
Arm/Group | CN + Combusted & Non-combusted Products | VLNC + Combusted & Non-combusted Products | VLNC With Non-combusted Products
Number analyzed (Participants) | 22 | 37 | 46
combuster products per day | 19.2 (8.1) | 12.9 (7.6) | 13.5 (9.8)

3. Secondary Outcome: Rate of 24 Hour Quit Attempts
Description: Rate of 24 hour quit attempts during the intervention period
Time Frame: 8 week intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | CN + Combusted & Non-combusted Products | VLNC + Combusted & Non-combusted Products | VLNC With Non-combusted Products
Number analyzed (Participants) | 27 | 53 | 56
Participants | 2 | 12 | 15

4. Secondary Outcome: Carcinogen Exposure Biomarker: Total NNAL
Description: Total NNAL (pmol/mg creatinine) is a measure of carcinogen exposure assessed at the end of intervention.
Time Frame: Week 8 (end of intervention)
Measure: Mean (95% Confidence Interval); unit: pmol//mg creatinine
Arm/Group | CN + Combusted & Non-combusted Products | VLNC + Combusted & Non-combusted Products | VLNC With Non-combusted Products
Number analyzed (Participants) | 22 | 37 | 46
pmol//mg creatinine | 1.22 [0.91 to 1.65] | 0.71 [0.41 to 1.23] | 0.51 [0.35 to 0.74]

ADVERSE EVENTS:
Time Frame: During the 8 week intervention
Arm/Group | CN + Combusted & Non-combusted Products | VLNC + Combusted & Non-combusted Products | VLNC With Non-combusted Products
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/53 | 1/56
Other Adverse Events (participants affected / at risk) | 6/27 | 7/53 | 23/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CN + Combusted & Non-combusted Products (N=27) | VLNC + Combusted & Non-combusted Products (N=53) | VLNC With Non-combusted Products (N=56)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Pneumonia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CN + Combusted & Non-combusted Products (N=27) | VLNC + Combusted & Non-combusted Products (N=53) | VLNC With Non-combusted Products (N=56)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 8 (8)
Headache (General disorders) | 0 (0) | 7 (7) | 5 (5)
Irritability (General disorders) | 2 (2) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Sore throat (General disorders) | 0 (0) | 0 (0) | 7 (7)
Difficulty concentrating (General disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Exploratory study due to small number of participants. Only used first generation of electronic cigarette products.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No